CLINICAL TRIAL: NCT02570061
Title: Recruiting to Clinical Trials on the Telephone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gorm Greisen (Other)
Responsible Party: Sponsor-Investigator, Gorm Greisen, consultant, professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H-4-2013 FSP-044
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Parental Consent; Newborn; Vaccination
Keywords: recruitment; comprehension; satisfaction; informed consent; telephone
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telephone (Experimental): Information about the Calmette study was given by telephone
  Interventions: Behavioral: telephone
- face-to-face (Active Comparator): Information about the Calmette study was given face-to-face at a consultation at the hospital
  Interventions: Behavioral: consultation face-to-face

INTERVENTIONS:
Behavioral: telephone — information given at the primary contact by phone, or at a scheduled later time
  Arms: telephone
Behavioral: consultation face-to-face — information given at a scheduled consultation at the hospital
  Arms: face-to-face

SUMMARY:
This study examined the use of the telephone for the purpose of informing expectant mothers about a randomized clinical trial assessing neonatal Bacille Calmette-Guérin vaccination. Expectant mothers who were contacted for participation in a vaccination trial (the Calmette study, NCT01694108) were randomized to receive information by telephone or at a face-to-face consultation. The primary outcome was a communication score, consisting of comprehension of information about the study and satisfaction with the information process. The outcome was measured using a questionnaire two weeks after the information was provided and two and a half months after birth.

DETAILED DESCRIPTION:
Informed consent is an essential element of clinical research. Obtaining consent, however, may be challenging. The use of the telephone for giving information and obtaining consent may be practical but little formal research has been done.

This study examined the use of the telephone for the purpose of informing expectant mothers about a randomized clinical trial assessing neonatal Bacille Calmette-Guérin vaccination. Expectant mothers who were contacted for participation in the Calmette Study were randomised to receive information by telephone or at a face-to-face consultation. The primary outcome was a communication score, consisting of comprehension of information about the study and satisfaction with the information process. The outcome was measured using a questionnaire two days after the information was provided and two and a half months after birth.

ELIGIBILITY:
Inclusion Criteria:

* Planning to give birth at Rigshospitalet

Exclusion Criteria:

* Prior contact to the Calmette trial staff
* Unable/unwilling to come to hospital for face-to-face information
* Declining participation in this trial

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
total communication score | 2 weeks after information was given
  Sum of scores of answers to all questions in a proprietary questionnaire

SECONDARY OUTCOMES:
comprehension subscore | 2 weeks after information was given
  comprehension of trial-related information: sum of scores of answers
satisfaction subscore | 2 weeks after information was given
  satisfaction with information process: sum of scores of answers
comprehension subscore | 2.5 months after birth of the infant
  comprehension of trial-related information: sum of scores of answers
satisfaction subscore | 2.5 months after birth of the infant
  satisfaction with information process: sum of scores of answers

CONTACTS AND LOCATIONS:
Overall Officials: Kim Foss, MD, Principal Investigator — Rigshospitalet, Denmark

REFERENCES:
- [Background] Thostesen LM, Nissen TN, Kjaergaard J, Pihl GT, Birk NM, Benn CS, Greisen G, Kofoed PE, Pryds O, Ravn H, Jeppesen DL, Aaby P, Stensballe LG. Bacillus Calmette-Guerin immunisation at birth and morbidity among Danish children: A prospective, randomised, clinical trial. Contemp Clin Trials. 2015 May;42:213-8. doi: 10.1016/j.cct.2015.04.006. Epub 2015 Apr 18. PMID 25896113
- [Derived] Foss KT, Kjaergaard J, Stensballe LG, Greisen G. Recruiting to Clinical Trials on the Telephone - a randomized controlled trial. Trials. 2016 Nov 21;17(1):552. doi: 10.1186/s13063-016-1680-y. PMID 27871308